CLINICAL TRIAL: NCT03825757
Title: Aggravated Airway Inflammation: Research on Genomics and Optimal Medical Care (AirGOs-medical)
Acronym: AirGOs-med
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanna Salmi (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Sanna Salmi, Senior Consultant Otorhinolaryngologist, PI, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYH2018203; 2017-001570-42 (EudraCT Number)
Record Dates: First submitted 2019-01-26; First posted 2019-01-31 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: chronic rhinosinusitis with nasal polyps; Acetyl salicylic acid exacerbated respiratory disease
MeSH Terms: conditions — Disease | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded controlled trial
Who Masked: Care Provider
Masking Description: The IMP producer (Galena Pharma Ltd., Kuopio, Finland) has packed the IMP according to study protocol and provides a code of each product. The IMP is used double-blinded in their numbered order. The key of the codes are stored in closed envelopes in Hospital´s locked closet. HYKS-institute performs regular study monitoring
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primaspan tablet 250 mg (Experimental): Primaspan tablet 250 mg (Acetyl salicylic acid): 1/2 tablet once daily during 1 month. 1 tablet once daily during 10 months. If not tolerated the dose 1 tablet x1/day, the patient is allowed to continue with the dose of 1/2 tablet x1/day.
  Interventions: Drug: Acetyl Salicylic Acid
- Placebo tablet (Placebo Comparator): Placebo Oral Tablet: 1/2 tablet once daily during 1 month. 1 tablet once daily during 10 months. If not tolerated the dose 1 tablet x1/day, the patient is allowed to continue with the dose of 1/2 tablet x1/day.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Placebo Oral Tablet — Placebo Oral Tablet
  Other Names: Placebo
  Arms: Placebo tablet
Drug: Acetyl Salicylic Acid — Primaspan 250 mg tablet Acetyl Salicylic Acid
  Other Names: Primaspan 250 mg tablet
  Arms: Primaspan tablet 250 mg

SUMMARY:
The study is performed as a randomized double-blinded prospective controlled trial. A total of 72 adult Acetyl salicylic acid (ASA) -exacerbated respiratory disease (AERD) -patients with uncontrolled chronic rhinosinusitis with nasal polyps (CRSwNP) will be recruited. Those negative to ASA-challenge test will not enter the Clinical Trial . All patients entering the Clinical Trial, have undergone earlier ethmoidal surgery (partial/total) and have not gained disease control. F-helicobacter antigen is tested and treatment is given if indicated. The patients are recruited at the Helsinki University Hospital (HUH). The study will be monitored by a professional monitor. Electronic CRF and paper/electronic patient questionnaires provided by HUS will be used (eCRF and patient questionnairea, Granitics).

DETAILED DESCRIPTION:
Randomization and the treatment arms I-II: The patients are randomized to two treatment arms I) ASA- desensitization po tablet daily for 11 months (n=36) II) Placebo po tablet daily for 11 months (n=18).

ASA challenge and desensitization (Primaspan) /Placebo: is conducted according to modified international protocol. FEV1 should be at least 1.5 L and > 60% of predicted before challenge or desensitization. On the first day every patient will receive 25 mg + 25 mg ASA at a hospital setting. On the second day every patient will receive 50 mg + 25 mg ASA at a hospital setting. On the third day every patient will receive 75 mg + 25 mg ASA at a hospital setting. On the fourth day every patient will receive 100 mg + 25 mg ASA at a hospital setting.

During the ASA challenge, patient who is ASA-challenge positive is then randomized and starts the trial so that he/she uses blinded ½ tablet of 250 mg ASA or ½ tablet of placebo daily at home for the next 1 month. After this period of 1 month, the dosing is increased at hospital setting, so that the patient receives blindly 250 mg ASA 1/2 tablet + 1/2 tablet or placebo 1/2 tablet + 1/2 tablet. Thereafter he/she will continue using blindly 250 mg ASA 1 tablet or placebo 1 tablet daily at home for the next 10 months. If the patient does not tolerate the up-dosing of ASA/placebo, he/she will continue using blindly ½ tablet of 250 mg ASA/placebo daily at home for the next 10 months. The total duration of the ASA/placebo treatment is 11 months. We additionally take nasal, blood and urine samples during the trial.

Follow-ups. The symptom questionnaire and interview of side-effects are performed during each visit. Lung function (eNO, nNO, PEF, spirometry) is monitored and the patient will visit doctor and/or nurse at 1, 5, 11, and 12 months post-starting with the treatment. Samples are taken during recruitment visit, before and after ASA-challenge and at 5, 11 and 12 months post-starting with the treatment. We also monitor side-effects, exacerbations, need of medication (po. cortisocteroids; antibiotics) and satisfaction to treatment.

Primary end point is change in nasal endoscopic nasal polyp score at -4 days vs. +11 months post-randomization. Secondary end point is change in Sinonasal Outcome Test -22 (SNOT-22) score at -4 days vs. +11 months post-randomization, and change in relative Forced expiratory volume in 1 second (FEV1 %) without bronchodilator at -1 month vs. +11 months post-randomization.

Safety (complications, adverse effects), costs and loss of productivity between study arms will be compared.

Trial medication will be discontinued, if surgery is needed before the end of follow-up.

ELIGIBILITY:
Inclusion Criteria: ALL these need to be positive:

* Endoscopic nasal polyp score ≥4
* SNOT-22 ≥30
* Sinus Computed tomography Lund-Mackay score ≥14. The new sinus CT scans are needed if the previous sinus CT scans have been performed over 36 months before recruitment visit or if there is a suspicion of complication of CRS (f.ex. mucocele, invasive fungal rhinosinusitis)
* ≥1 previous partial/total ethmoidectomy surgery.

In addition, patient should have a history of at least one of the following:

>1 oral corticosteroids during the past two years >3 antibiotic courses during the past two years. In patients with contraindication/adverse effects in using oral steroids additional criteria are not required.

Exclusion Criteria:

* complication of CRS (f.e. mucocele, invasive fungal rhinosinusitis)
* bleeding diathesis
* pregnancy/ breastfeeding
* cystic fibrosis
* primary ciliary dyskinesia (PCD)
* sarcoidosis
* granulomatosis with polyangitis (GPA)
* eosinophilic granulomatosis with polyangitis (EGPA)
* immunosuppression (diagnosed Spesific antibody deficiency (SAD), CVI, HIV
* use of biologicals/immunosuppressive medication
* immunotherapy
* Daily use of systemic corticosteroids (Prednisolon 10mg or equivalent) -communication problems (f.e. neurological/psychiatric disease, language skills) -unlikely to comply
* other severe disease
* uncontrolled asthma
* ASA-challenge negative
* gastric ulcer
* anticoagulant treatment
* SSRI-depression medication
* beta-blocker
* severe chronic urticaria
* ASA anaphylaxis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Change in endoscopic Nasal polyp score of both sides of the nasal cavity. | at -4 days vs. at 11 months post-randomization
  Change means differences between at time -4 days versus (vs.) at time +11 months post-randomization. Minimum value is 0. Maximum value is 8. A higher score means worse outcome.

SECONDARY OUTCOMES:
Change in Sinonasal outcome test 22 (SNOT22). Validated nose-specific quality of life questionnaire, 0-110 points. | at -4 days vs. at 11 months post-randomization
  Change means differences between at time -4 days vs. +11 months post-randomization. A higher score means worse outcome.
Change in the Relative forced expiratory volume in 1 second (FEV1%) without bronchodilator. | at -1 month vs. at 11 months post-randomization
  Change means differences between at time -1 month vs. +11 months post-randomization. A higher value means better outcome. FEV1% is measured by Spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Sanna Toppila-Salmi, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
The data is owned by Helsinki University Hospital and University of Helsinki.

REFERENCES:
- [Derived] Toppila-Salmi S, Lyly A, Salmi V, Nuutinen M, Kilpio M, Hanif T, Niemi M, Laulajainen-Hongisto A, Hafren L, Makela M, Kauppi P, Virkkula P, Heleva A. Study protocol for a randomized double-blinded placebo-controlled trial on ASA therapy for patients with chronic rhinosinusitis with nasal polyps, NSAID-exacerbated respiratory disease, and asthma. Front Allergy. 2025 May 20;6:1542481. doi: 10.3389/falgy.2025.1542481. eCollection 2025. PMID 40463360
- See also: Diagnosis and management of NSAID-Exacerbated Respiratory Disease (N-ERD)-a EAACI position paper. — https://www.ncbi.nlm.nih.gov/pubmed/30216468
- See also: Aspirin-Exacerbated Respiratory Disease. Publication. — https://www.ncbi.nlm.nih.gov/pubmed/30575459